CLINICAL TRIAL: NCT01451775
Title: Investigation of the Effect of Food on the Bioavailability of a 25 mg Empagliflozin Tablet and Assessment of Dose Proportionality Between 10 mg and 25 mg Empagliflozin Tablets in an Open, Randomised, Single Dose, Three-period Cross-over Study in Healthy Male and Female Subjects
Brief Title: Investigation of the Effect of Food on the Bioavailability of a 25 mg Empagliflozin Tablet as Well as Assessment of Dose Proportionality Between 10 mg and 25 mg Empagliflozin Tablets Under Fasting Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.79; 2011-002836-13 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (3):
- Treatment A (Experimental): high dose of empagliflozin after overnight fasting for at least 10 h
  Interventions: Drug: Empagliflozin
- Treatment B (Experimental): high dose of empagliflozin after a standardised high fat breakfast
  Interventions: Drug: Empagliflozin
- Treatment C (Experimental): low dose empagliflozin after overnight fasting for at least 10 h
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — high dose of empagliflozin after overnight fasting for at least 10 h
  Arms: Treatment A
Drug: Empagliflozin — low dose empagliflozin after overnight fasting for at least 10 h
  Arms: Treatment C
Drug: Empagliflozin — high dose of empagliflozin after a standardised high fat breakfast
  Arms: Treatment B

SUMMARY:
Investigation of food effect on the bioavailability of a 25 mg empagliflozin tablet and assessment of dose proportionality between 10 mg and 25 mg empagliflozin tablets under fasting conditions.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.79.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised 3 period crossover trial. 18 patients were randomised to one of six treatment sequences and treated. The trial was open label with washout periods of at least 7 days between treatments.
Groups:
- Empa 25mg Fasted / Empa 25mg Fed / Empa 10mg Fasted: Patients were administered three treatments in the following order:
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
- Empa 25mg Fasted / Empa 10mg Fasted / Empa 25mg Fed: Patients were administered three treatments in the following order:
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
- Empa 25mg Fed / Empa 25mg Fasted / Empa 10mg Fasted: Patients were administered three treatments in the following order:
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
- Empa 25mg Fed / Empa 10mg Fasted / Empa 25mg Fasted: Patients were administered three treatments in the following order:
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
- Empa 10mg Fasted / Empa 25mg Fasted / Empa 25mg Fed: Patients were administered three treatments in the following order:
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
- Empa 10mg Fasted / Empa 25mg Fed / Empa 25mg Fasted: Patients were administered three treatments in the following order:
  * A single dose of 10 mg empa after an overnight fast of at least 10 hours.
  * A single dose of 25 mg empa after a standardised high-fat, high-caloric breakfast
  * A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Empa 25mg Fasted / Empa 25mg Fed / Empa 10mg Fasted | Empa 25mg Fasted / Empa 10mg Fasted / Empa 25mg Fed | Empa 25mg Fed / Empa 25mg Fasted / Empa 10mg Fasted | Empa 25mg Fed / Empa 10mg Fasted / Empa 25mg Fasted | Empa 10mg Fasted / Empa 25mg Fasted / Empa 25mg Fed | Empa 10mg Fasted / Empa 25mg Fed / Empa 25mg Fasted
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: Total number of patients randomised and treated in the study. This was a randomised 3 period crossover trial. 18 patients were randomised to one of six treatment sequences and treated. The trial was open label with washout periods of at least 7 days between treatments.
Arm/Group | Study Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 hours extrapolated to infinity (AUC0-∞).
  The Measured Values show intra-arm variabilities, whereas the statistical analyses show inter-arm variabilities.
Time Frame: 1 hour (h) before study drug and 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: All treated subjects who provided at least one observation in the relevant treatment periods for at least one primary pharmacokinetic (PK) endpoint without a relevant protocol deviation and who had not experienced emesis before or at 2 times median tmax in at least one of the two relevant treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa 25 mg Fasted: A single dose of 25 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
- Empa 25 mg Fed: A single dose of 25 mg empagliflozin (empa) after a standardised high-fat, high-caloric breakfast.
- Empa 10 mg Fasted: A single dose of 10 mg empagliflozin (empa) after an overnight fast of at least 10 hours.
Arm/Group | Empa 25 mg Fasted | Empa 25 mg Fed | Empa 10 mg Fasted
Number analyzed (Participants) | 18 | 17 | 18
nmol*h/L | 5380 (26.0) | 4520 (24.8) | 2280 (27.0)
Statistical Analysis 1: Comparison: Empa 25 mg Fasted vs Empa 25 mg Fed; Test type: Non-Inferiority or Equivalence — Bioavailability study with standard bioequivalence range of 80% to 125%. Ratio calculated as empa 25mg fed divided by empa 25mg fasted; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 84.04, 90% CI 2-sided [80.856 to 87.344], Standard Deviation 6.4 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Empa 25 mg Fasted vs Empa 10 mg Fasted; Test type: Non-Inferiority or Equivalence — This is an analysis of dose proportionality; ANCOVA — Does proportionality would be assumed if the 95% confidence interval includes one; ANCOVA with logarithm of the dose fitted as a continuous covariate and sequence, subjects within sequence, period included as categorical variables; Slope = 0.9367, 95% CI 2-sided [0.8988 to 0.9746], Standard Error of Mean 0.0178

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagloflozin (empa) in plasma, per period.
  The Measured Values show intra-arm variabilities, whereas the statistical analyses show inter-arm variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa 25 mg Fasted | Empa 25 mg Fed | Empa 10 mg Fasted
Number analyzed (Participants) | 18 | 17 | 18
nmol/L | 837 (27.8) | 523 (27.7) | 365 (27.7)
Statistical Analysis 1: Comparison: Empa 25 mg Fasted vs Empa 25 mg Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 63.22, 90% CI 2-sided [56.736 to 70.439], Standard Deviation 18.1 — Standard deviation is actually the geometric coefficient of variation
Statistical Analysis 2: Comparison: Empa 25 mg Fasted vs Empa 10 mg Fasted; Test type: Non-Inferiority or Equivalence — This is an analysis of dose proportionality; ANCOVA — Does proportionality would be assumed if the 95% confidence interval includes one; [statistical method as in outcome 1, analysis 2]; Slope = 0.9065, 95% CI 2-sided [0.8011 to 1.0120], Standard Deviation 0.0495

3. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Clinical Laboratory Tests and Assessment of Tolerability by the Investigator.
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, blood chemistry, haematology, urinanalysis and assessment of tolerability by the investigator. New abnormal findings or worsening of baseline conditions were reported as adverse events (AEs). Time frame for AE reporting includes the period of first drug administration until end of study. A more detailed definition of the used time frame and MedDRA Version can be found in the AE section.
Time Frame: Screening until end of trial, average of 45 days
Population: Treated Set(TS): TS includes all subjects who have taken at least 1 dose of trial medication
Measure: Number; unit: participants
Arm/Group | Empa 25 mg Fasted | Empa 25 mg Fed | Empa 10 mg Fasted
Number analyzed (Participants) | 18 | 18 | 18
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Drug administration until beginning of next sequence/end of trial, average of 24 days
Arm/Group | Empa 25 mg Fasted | Empa 25 mg Fed | Empa 10 mg Fasted
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 2/18 | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 25 mg Fasted (N=18) | Empa 25 mg Fed (N=18) | Empa 10 mg Fasted (N=18)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes